CLINICAL TRIAL: NCT05138874
Title: Improving Safe Antibiotic Prescribing in Telehealth: Evaluation of a Randomized Trial
Brief Title: Improving Safe Antibiotic Prescribing in Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Teladoc Health (Industry)
Responsible Party: Principal Investigator, Daniella Meeker, Associate Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01HS026506 (AHRQ)
Record Dates: First submitted 2021-10-20; First posted 2021-12-01 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Infection; Telehealth
Keywords: antibiotics; behavioral economics; social norms; performance feedback

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three levels of commitment interventions and one of three levels of feedback interventions, for a total of 9 study arms (3 X 3). One level in each factor is "control" which entails "no intervention".
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients are blinded to all study arms with the exception of Public Commitment where, by design, patients are exposed to physicians' commitment. Physicians cannot be blinded to interventions that, by design, impact the electronic medical record display.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Trending Feedback + Private Commitment (Experimental): Clinicians receive both Trending Feedback + Private Commitment interventions.
  Interventions: Behavioral: Trending Feedback; Behavioral: Private Commitment
- Trending Feedback + Public Commitment (Experimental): Clinicians receive both Trending Feedback + Public Commitment interventions.
  Interventions: Behavioral: Trending Feedback; Behavioral: Public Commitment
- Trending Feedback + Commitment Control (Experimental): Clinicians receive Trending Feedback intervention + Commitment Control.
  Interventions: Behavioral: Trending Feedback
- Benchmark Peer Comparison Feedback + Private Commitment (Experimental): Clinicians receive both Benchmark Peer Comparison Feedback + Private Commitment interventions.
  Interventions: Behavioral: Benchmark Peer Comparison Feedback; Behavioral: Private Commitment
- Benchmark Peer Comparison Feedback + Public Commitment (Experimental): Clinicians receive both Benchmark Peer Comparison Feedback + Public Commitment interventions.
  Interventions: Behavioral: Benchmark Peer Comparison Feedback; Behavioral: Public Commitment
- Benchmark Peer Comparison Feedback + Commitment Control (Experimental): Clinicians receive Benchmark Peer Comparison Feedback intervention + Commitment Control.
  Interventions: Behavioral: Benchmark Peer Comparison Feedback
- Public Commitment + Feedback Control (Experimental): Clinicians receive Public Commitment intervention + Feedback Control.
  Interventions: Behavioral: Public Commitment
- Private Commitment + Feedback Control (Experimental): Clinicians receive Private Commitment intervention + Feedback Control.
  Interventions: Behavioral: Private Commitment
- Commitment Control + Feedback Control (No Intervention): Clinicians receive no intervention.

INTERVENTIONS:
Behavioral: Trending Feedback — Clinicians randomized to Trending Feedback will receive monthly feedback on the provider dashboard page.
  Arms: Trending Feedback + Commitment Control; Trending Feedback + Private Commitment; Trending Feedback + Public Commitment
Behavioral: Benchmark Peer Comparison Feedback — Clinicians randomized to Benchmark Peer Comparison Feedback will receive monthly feedback on the provider dashboard page.
  Arms: Benchmark Peer Comparison Feedback + Commitment Control; Benchmark Peer Comparison Feedback + Private Commitment; Benchmark Peer Comparison Feedback + Public Commitment
Behavioral: Private Commitment — Clinicians assigned to the Private Commitment will be prompted in the provider dashboard to make a personal commitment to evidence-based use of antibiotics that will not be shared with their patients.
  Arms: Benchmark Peer Comparison Feedback + Private Commitment; Private Commitment + Feedback Control; Trending Feedback + Private Commitment
Behavioral: Public Commitment — Clinicians assigned to Public Commitment will be prompted in the provider dashboard to make a commitment to evidence-based use of antibiotics that will be shared with their patients.
  Arms: Benchmark Peer Comparison Feedback + Public Commitment; Public Commitment + Feedback Control; Trending Feedback + Public Commitment

SUMMARY:
Appropriate use of antibiotics reduces resistance and protects patients from unnecessary harm. Important advances in antibiotic stewardship have been achieved in outpatient settings, but little is known about stewardship in the rapidly growing telehealth sector. Prior pragmatic randomized trials have shown that Centers for Disease Control (CDC) Core Element interventions constructed using insights from decision and social psychology can greatly reduce inappropriate prescribing in outpatient settings.

In a randomized trial, the investigators will adapt and test two aspects of CDC Core Elements in a telehealth environment (Teladoc®), each with two levels of intensity. Teladoc® clinicians will be randomized to the following interventions: 1) Performance Feedback (Trending, Benchmark Peer Comparison), 2) Commitment (Private, Public), or 3) Control. All randomization occurs at the provider level, with the exception of the Public Commitment arm, which requires patient-facing content that is determined by patient state. Clinicians and members will see the same messages across all pages, all channels & all consults during the 12-month study period. The primary outcome is to assess change in antibiotic prescribing rate for qualifying acute respiratory infection visits (ARIs).

DETAILED DESCRIPTION:
In a 3 x 3 (Performance Feedback x Commitment) randomized trial, the investigators will adapt and test two aspects of Core Elements in a telehealth environment (Teladoc®), each with two variations. Qualifying visits include pediatric and adult telehealth visits for acute respiratory infections, including sinusitis, bronchitis, influenza, otitis media, pharyngitis, nonspecific upper respiratory infections, and COVID-19.

All randomization occurs at the provider level, with the exception of the Public Commitment arm, which requires patient-facing content that is determined by patient state. Allocation will be stratified to ensure balance across baseline characteristics including visit volume (consults per year), antibiotic prescribing rate for acute respiratory infections and COVID-19, and average member satisfaction (percent of responses "Outstanding" or "Good").

Performance Feedback (Trending, Benchmark Peer Comparison, Control). Performance Feedback is based on regional performance benchmarks; physicians with antibiotic prescribing rates in the lowest 3 deciles are designated top performers. The electronic health record (EHR) metrics and messaging are designed to align with enterprise-wide performance feedback practices. A minimum of 8 qualifying visits is required for a provider to see a message.

Providers randomized to Performance Feedback interventions will see one of two feedback messages in the EHR:

1. Trending Feedback Message: If the clinician's mean monthly antibiotic prescribing rate for acute respiratory infections is below the 3rd decile, where better performance is indicated by a position in a lower decile, providers will see the following message with a link to the clinical practice guidelines: "Your antibiotic prescribing rate is X%. Stay in the growing number of providers in your group that have stopped inappropriate antibiotic prescribing." If the clinician's mean monthly antibiotic prescribing rate for ARIs is above the 3rd decile where better performance is indicated by a position in a lower decile, providers will see the following message with a link to the clinical practice guidelines: "Your antibiotic prescribing rate is Y% (where Y% is the prescribing rate of the third decile). Don't be left behind! Join the growing number of providers in your group who prescribe antibiotics only when clearly indicated."
2. Benchmark Peer Comparison Feedback Message: If the clinician's mean monthly antibiotic prescribing rate for ARIs is below the 3rd decile, where better performance is indicated by a position in a lower decile, providers will receive the following message: "You are a Top Performer. Your antibiotic prescribing rate is X%. Top performers in your group typically prescribe antibiotics in X% of visits." If the clinician prescribing rate is above the 3rd decile, where better performance is indicated by a position in a lower decile, providers will receive the following message: "You are not a Top Performer. Top performers in your group typically prescribe antibiotics in Y% of visits."

Commitment (Private, Public, Control). Clinicians assigned to the Private Commitment arm will make a personal commitment to evidence-based use of antibiotics that is not shared with their patients, while those assigned to Public Commitment will make a commitment to evidence-based use of antibiotics that is shared with their patients. For both arms, this commitment is displayed on the clinician's personal provider dashboard.

Providers randomized to the Commitment interventions will be asked to complete one of two commitments:

1. Private Commitment: Providers will be given the following options:1) Record my commitment or 2) Do not include me in the commitment, followed by a text box to type their name. For clinicians who choose option 1, their commitment is displayed on their personal provider dashboard at the time of each login.
2. Public Commitment: Providers will be given the following options:1) Record and share my commitment with my patients OR 2) I am not committed to the new guidelines, followed by a text box to type their name. For clinicians who opt in, the commitment is displayed on their personal dashboard at each login.

Patients in states assigned to Public Commitment will see the clinician's commitment at the end of their visit request. Patients will select: 1) I understand the provider's commitment OR 2) I do not understand and need more information. Clinicians in this arm will be notified about the patient response in the EHR during the visit.

The primary outcome is to assess the change in antibiotic prescribing rate for qualifying acute respiratory infection visits.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians with prescribing privileges and one or more Acute Respiratory Infection visit
* Eligible encounters include pediatric and adult telehealth visits for Acute Respiratory Infections, including Sinusitis, Bronchitis, Influenza, Otitis Media, Nasopharyngitis, Upper Respiratory Infections, and COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6581 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Change in antibiotic prescribing rate for Acute Respiratory Infections | 12 months
  Change in antibiotic prescribing rate for acute respiratory infection visits based on the International Statistical Classification of Diseases, version 10 (ICD-10) codes including: non-specific upper respiratory infections, otitis media, sinusitis, pharyngitis, bronchitis, influenza, and COVID-19.

SECONDARY OUTCOMES:
Change in inappropriate antibiotic prescribing rate for Acute Respiratory Infections | 12 months
  Change in inappropriate antibiotic prescribing rate for acute respiratory infections where antibiotics are never appropriate based on International Statistical Classification of Diseases, version 10 (ICD-10) codes as well as COVID-19 (U07.1)

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Meeker, PhD, Principal Investigator — University of Southern California
Locations (1):
- Teladoc Health, Dallas, Texas, United States

REFERENCES:
- [Background] Chua KP, Fischer MA, Linder JA. Appropriateness of outpatient antibiotic prescribing among privately insured US patients: ICD-10-CM based cross sectional study. BMJ. 2019 Jan 16;364:k5092. doi: 10.1136/bmj.k5092. PMID 30651273
- [Background] Meeker D, Knight TK, Friedberg MW, Linder JA, Goldstein NJ, Fox CR, Rothfeld A, Diaz G, Doctor JN. Nudging guideline-concordant antibiotic prescribing: a randomized clinical trial. JAMA Intern Med. 2014 Mar;174(3):425-31. doi: 10.1001/jamainternmed.2013.14191. PMID 24474434
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- [Background] Sanchez GV, Fleming-Dutra KE, Roberts RM, Hicks LA. Core Elements of Outpatient Antibiotic Stewardship. MMWR Recomm Rep. 2016 Nov 11;65(6):1-12. doi: 10.15585/mmwr.rr6506a1. PMID 27832047
- [Background] Linder JA, Meeker D, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Doctor JN. Effects of Behavioral Interventions on Inappropriate Antibiotic Prescribing in Primary Care 12 Months After Stopping Interventions. JAMA. 2017 Oct 10;318(14):1391-1392. doi: 10.1001/jama.2017.11152. PMID 29049577
- [Derived] McCabe BK, Linder JA, Doctor JN, Friedberg M, Fox CR, Goldstein NJ, Knight TK, Kaiser K, Tibbels J, Haenchen S, Persell SD, Warberg R, Meeker D. The protocol of improving safe antibiotic prescribing in telehealth: A randomized trial. Contemp Clin Trials. 2022 Aug;119:106834. doi: 10.1016/j.cct.2022.106834. Epub 2022 Jun 18. PMID 35724841